CLINICAL TRIAL: NCT06043687
Title: Clinical Efficacy of Two Different Dentifrice Formulations in Treatment of Chronic Periodontitis
Brief Title: Efficacy of Herbal Dentifrice in Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Collaborators: Jasberry Healthcare Pvt. Ltd (Unknown)
Responsible Party: Principal Investigator, D. Gopalakrishnan, Dean, Professor and HOD, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DYPV/EC/883/22/B
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dentifrice containing Jasmate formulation (Experimental): Patients will be instructed to brush twice daily. Patients will be instructed to apply at least a 1-inch strip of the Jasmate formulation toothpaste onto a soft toothbrush and to brush thoroughly for 2 minutes and expectorate. All patients will be instructed to use only the assigned products and refrain from other dentifrice or mouth-rinse during the trial but will be allowed to continue their normal oral hygiene practices. Patients will use the assigned product for a period of 24 weeks for assessment of the efficacy and safety in periodontitis patients.
  Interventions: Drug: Dentifrice Paste
- Dentifrice containing Biomin formulation (Active Comparator): Patients will be instructed to brush twice daily. Patients will be instructed to apply at least a 1-inch strip of the Biomin formulation toothpaste onto a soft toothbrush and to brush thoroughly for 2 minutes and expectorate. All patients will be instructed to use only the assigned products and refrain from other dentifrice or mouth-rinse during the trial but will be allowed to continue their normal oral hygiene practices. Patients will use the assigned product for a period of 24 weeks for assessment of the efficacy and safety in periodontitis patients.
  Interventions: Drug: Dentifrice Paste
- Dentifrice containing placebo formulation (Placebo Comparator): Patients will be instructed to brush twice daily. Patients will be instructed to apply at least a 1-inch strip of the Placebo formulation toothpaste onto a soft toothbrush and to brush thoroughly for 2 minutes and expectorate. All patients will be instructed to use only the assigned products and refrain from other dentifrice or mouth-rinse during the trial but will be allowed to continue their normal oral hygiene practices. Patients will use the assigned product for a period of 24 weeks for assessment of the efficacy and safety in periodontitis patients.
  Interventions: Drug: Dentifrice Paste

INTERVENTIONS:
Drug: Dentifrice Paste — Scaling and Root planing followed by dentifrice usage

SUMMARY:
The study will be a single center, longitudinal prospective, triple blind (investigators, patients and statistician), randomized design. After informed consent, a target population of about 75 healthy adult volunteers with periodontitis will be included in the study. Patients will be randomized and categorized into three experimental groups each containing 25 patients. The randomization process will be carried out by use of sequentially numbered opaque sealed envelopes (SNOSE method).The recording of all the soft tissues data plaque index, gingival index, the modified sulcus bleeding index and the periodontal probing depth and clinical attachment level will be carried out at baseline, 4 weeks, 8 weeks, 12 weeks and will be maintained till 24 weeks for efficacy and safety evaluation.

DETAILED DESCRIPTION:
Patients will be instructed to brush twice daily. Patients will be instructed to apply at least a 1-inch strip of the toothpaste onto a soft toothbrush and to brush thoroughly for 2 minutes and expectorate. All patients will be instructed to use only the assigned products and refrain from other dentifrice or mouth-rinse during the trial but will be allowed to continue their normal oral hygiene practices. Patients will use the assigned product for a period of 24 weeks for assessment of the efficacy and safety in periodontitis patients.

A complete and detail oral examination will then be conducted to evaluate the oral and perioral region, including soft tissues. Patients will return at study location at 4 weeks, 8 weeks, 12 weeks and 24 weeks for the soft-tissue assessment using the plaque index, gingival index, the modified sulcus bleeding index and the periodontal probing depth and clinical attachment level.

The following objectives will be assessed -

Objectives:

1. To assess efficacy and safety of Jasmate toothpaste preparation over a period of 24 weeks.
2. To evaluate the change in PI, GI, mSBI, PPD, CAL, in chronic periodontitis patients following scaling and root planing at 4 weeks, 8 weeks, 12 weeks and 24 weeks compared to baseline using Jasmate toothpaste preparation.
3. To evaluate the change in PI, GI, mSBI, PPD, CAL, in chronic periodontitis patients following scaling and root planing at 4 weeks, 8 weeks, 12 weeks and 24 weeks compared to baseline using BioMin Ftoothpaste preparation.
4. To compare the change in PI, GI, mSBI, PPD, CAL in chronic periodontitis patients following scaling and root planing at 4 weeks, 8 weeks, 12 weeks and 24 weeks using Jasmate toothpaste preparation and BioMin Ftoothpaste preparation.

ELIGIBILITY:
Inclusion Criteria:

* The patient should be in good general health as determined by the Investigator/ medical expert;
* The patient should agree not to participate in any other oral/dental product studies during the course of this study;
* The patient should agree to delay any dental treatment until the study has been completed;
* The patient should agree to abstain from the use of any non-study oral hygiene products;
* The patient should exhibit adequate oral hygiene (i.e., brush teeth daily and exhibit no signs of oral neglect);
* The patient should agree to return for all scheduled visits and follow study procedures;
* The patient should have a minimum of 20 teeth
* The periodontal status of the patient should be Mild to moderate periodontitis (AAP classification 1999)
* The oral status of the patient should be as follows:

Plaque index (Silness & Löe 1964)>2 Gingival Index (Löe and Silness 1963) >1.5 Modified Sulcus Bleeding Index (Mombelli et al 1987) >1 PPD > 4mm

Exclusion Criteria:

* Presence of any condition, abnormality or situation at baseline that in the opinion of the Principal Investigator may preclude the volunteer's ability to comply with study requirements, including completion of the study or the quality of the data
* Pregnant females
* Patients having history of Tobacco use
* Patients with Sjögren's disease
* Patients having immune deficiency diseases, i.e., HIV or AIDS
* Patients with poorly controlled diabetes mellitus
* Patients taking anti TNF-alpha medication for rheumatoid arthritis
* Patients taking anti-inflammatory, analgesic, or psychotropic drugs,
* Patients having self-reported eating disorders, uncontrolled gastroesophageal reflux disease (GERD or Acid Reflux), excessive dietary or environmental exposure to acids, or other systemic conditions that are predisposing to dentinal hypersensitivity;
* Patients with a history or presence of kidney disorders, kidney stones, celiac disease, inflammatory bowel disease (ulcerative colitis or Crohn's disease), chronic pancreatitis, have had intestinal or weight-loss surgery, or if have stomach or intestinal problems that keep them from absorbing certain foods or nutrients;
* The teeth will be excluded from study measurements if they have deep, defective, or facial restorations; have full crowns, extensive caries, cracked enamel, or are abutment teeth for fixed or removable prosthesis;
* The teeth having endo-perio lesion.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Clinical attachment level | Baseline to 24 weeks
  Change in Clinical attachment level in chronic periodontitis patients following scaling and root planing & dentifrice usage

SECONDARY OUTCOMES:
Change in Probing pocket depth | Baseline to 24 weeks
  Change in Probing pocket depth in chronic periodontitis patients following scaling and root planing & dentifrice usage
Change in Plaque Index levels | Baseline to 24 weeks
  Change in Plaque index levels in chronic periodontitis patients following scaling and root planing & dentifrice usage
Change in Gingival index levels | Baseline to 24 weeks
  Change in Gingival index levels in chronic periodontitis patients following scaling and root planing & dentifrice usage
Change in mean sulcus bleeding index levels | Baseline to 24 weeks
  Change in mean sulcus bleeding index levels in chronic periodontitis patients following scaling and root planing & dentifrice usage

CONTACTS AND LOCATIONS:
Overall Officials: Dharmarajan Gopalakrishnan, MDS, PhD, Principal Investigator — Dr. D Y Patil Dental College and Hospital, Pimpri, Pune
Locations (1):
- Dr. D Y Patil Dental College and Hospital, Pimpri, Pune, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No